CLINICAL TRIAL: NCT00925743
Title: A Dose-Escalation Study Of The Safety, Tolerability, And Pharmacokinetics Of Cabazitaxel In Combination With Cisplatin Administered Every 3 Weeks In Subjects With Advanced Solid Malignancies
Brief Title: A Study to Evaluate the Effects of Combining Cabazitaxel With Cisplatin Given Every 3 Weeks in Patients With Advanced Solid Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD10870
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Solid Cancer
Keywords: Phase 1; XRP6258; cisplatin; Antineoplastic Combined Chemotherapy Protocols
MeSH Terms: interventions — cabazitaxel; XRP6258

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): * 5, 15, 20 or 25 mg/m2
  * one injection of cabazitaxel on day 1 of each cycle (3 weeks)
  Interventions: Drug: cabazitaxel (XRP6258)

INTERVENTIONS:
Drug: cabazitaxel (XRP6258) — * administered by IV infusion
  * in addition to cisplatin treatment

SUMMARY:
This study is designed as a phase 1, multicenter, open-label, single arm, dose-escalation, study of Cabazitaxel in combination with cisplatin, to determine safety, pharmacokinetics (PK), and efficacy in solid tumors (parts 1 and 2) and single sequence, two-treatment, crossover studies to determine the effect of strong CYP3A4 inhibition and induction on the PK of Cabazitaxel in patients with solid tumors (part 3 and part 4, respectively).

There are 4 parts to the study:

Part 1: Determine the Dose Limiting Toxicities (DLT)'s and Maximum Tolerated Dose (MTD) based on safety.

Part 2: Determine the anti-tumor activity of the combination regimen at the Maximum Tolerated Dose (MTD) in an extended cohort of patients.

Part 3: Determine the effect of a strong CYP3A4 inhibitor (ketoconazole) on the pharmacokinetic (PK) of Cabazitaxel.

Part 4: Determine the effect of a strong CYP3A4 inducer (rifampin) on the pharmacokinetic (PK) of Cabazitaxel.

DETAILED DESCRIPTION:
The total duration on the study per subject will be about 26 weeks broken down as follows:

* A maximum of 21-day screening phase,
* 21-days (+/- 2 weeks) study treatment cycles,
* 30-day follow-up visit after the last dose of study medication.
* Cut-off date for parts 1, 2, 3 and 4: when the last patient has completed 6 cycles (parts 1 and 2) or 2 cycles (parts 3 and 4) of treatment or discontinued study treatment (for disease progression, unacceptable toxicity, withdrawal of consent, or investigator's decision to withdraw), whichever comes first, in the corresponding part.

Patients still receiving treatment at the cut-off date may continue to receive treatment beyond the cut-off date at investigator's discretion if benefiting.

ELIGIBILITY:
Inclusion criteria:

* confirmed metastatic or unremovable advanced solid malignancy that is metastatic or unresectable, and for which standard curative measures do not exist, but for which cisplatin based therapy is appropriate
* signed informed consent

Exclusion criteria

* limited physical functioning (as evaluated by the Eastern Cooperative Oncology Group (ECOG) scale)
* inability to follow study requirements and schedule
* treatment of cancer within 3 weeks of study, concurrent treatment in another clinical trial or with any other cancer therapy
* serious medical illness at same time of study and/or significantly abnormal lab reports
* lack of pregnancy contraception (women of childbearing potential), pregnancy, or breast feeding.
* Women of childbearing potential not protected by highly effective contraceptive method of birth control OTHER than hormonal contraception (Part 4 only).
* prior significant hearing or kidney problems
* continued toxic effects of prior chemotherapy
* cancers that cannot be physically measured (Part 2 only)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT)'s of the combination of cabazitaxel and cisplatin (part 1) | first cycle (i.e.3 weeks)
Objective response ratio (Complete response (CR) and partial response (PR)) (part 2) | up to 6 cycles, ie 18 weeks
Pharmacokinetics (PK) of cabazitaxel (part 3 and 4) | up to 6 cycles, ie 18 weeks

SECONDARY OUTCOMES:
Time to progression (TTP) (part 1 and 2) | up to 6 cycles, ie 18 weeks
Duration of response (DR) (Part 1 and 2) | up to 6 cycles, ie 18 weeks
Cabazitaxel pharmacokinetic (part 1 and 2) | up to 6 cycles, ie 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (7):
- United States (7):
  - Investigational Site Number 840008, Los Angeles, California
  - Investigational Site Number 840003, San Diego, California
  - Investigational Site Number 840010, Decatur, Illinois
  - Investigational Site Number 840002, Baltimore, Maryland
  - Investigational Site Number 840006, St Louis, Missouri
  - Investigational Site Number 840007, Cincinnati, Ohio
  - Investigational Site Number 840005, San Antonio, Texas

REFERENCES:
- [Derived] Lockhart AC, Sundaram S, Sarantopoulos J, Mita MM, Wang-Gillam A, Moseley JL, Barber SL, Lane AR, Wack C, Kassalow L, Dedieu JF, Mita AC. Phase I dose-escalation study of cabazitaxel administered in combination with cisplatin in patients with advanced solid tumors. Invest New Drugs. 2014 Dec;32(6):1236-45. doi: 10.1007/s10637-014-0145-y. Epub 2014 Aug 13. PMID 25117475